CLINICAL TRIAL: NCT01674920
Title: CHOICES: Family Physicians Treat Overweight Children
Acronym: CHOICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HD050962 (NIH); 1R21HD050962 (NIH)
Record Dates: First submitted 2008-05-18; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Obesity; Overweight
Keywords: Pediatric obesity; resiliency; physical activity; dietary patterns; children
MeSH Terms: conditions — Obesity; Overweight; Pediatric Obesity; Motor Activity | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Choices (Experimental): The 3-month twelve-session intervention, "Choices", included topics on nutrition, physical activity, and resiliency. Parents, boys and girls met separately. The sessions were developed for delivery by a family physician, two family medicine residents, and a nutritionist, who received training in positive psychology and resilience skills. All children were measured on the same dates, but children were randomly assigned to two cohorts, beginning 6 months apart, to facilitate statistical analysis by having one group experience "normal growth" on study prior to intervention.
  Interventions: Behavioral: Choices

INTERVENTIONS:
Behavioral: Choices — The 12-week intervention included 1.5 hour classes each week. Topics included nutrition, physical activity, and psychosocial skills based in Resiliency.
  Other Names: Resiliency; Nutrition; Physical Activity

SUMMARY:
CHOICES is a program to provide children and families with lifetime tools and lifestyle strategies to achieve and maintain a healthy body size. Both parents and children get active, learn about the food choices they can make, and about the roles of TV in their lives. Led by physicians and young adults, the 12 weekly 90 minute sessions provide hands on experiences that connect into the participants' daily lives. In the study, the families were divided into two groups, beginning their classes 6 months apart. Body measurements were taken at baseline and every 4 months to 16 months.

DETAILED DESCRIPTION:
The specific aim of this pilot study was to use the group office visit model to provide an obesity treatment intervention for children 8-11 years of age in gender-specific groups and their parents in a clinic setting. The targeted lifestyle components of the intervention are less TV viewing, less sweetened beverages, smaller food portions, less fast food/better choices away from home and more general physical activity. The psychosocial component was based in Resiliency; the Choices model focused on a non-judgmental approach to empowerment in relation to personal goals and knowledge of the basics of nutrition and physical activity.

Our aim was to recruit 35-40 children (approximately equal boys and girls) ages 8-11 and their parents for a 12 weekly sessions group office visit program. Participants were randomized into 2 groups; one group starting in March 2006 and the lagged intervention control group starting in September 2006. Physical measurements and data collection were at baseline, 4, 8, 12, 16 months from randomization.

We evaluated the acceptability and feasibility of the group office visit model and effect size (body mass index (BMI) and weight-for-age Z-scores). Feasibility and acceptability included ability to recruit within clinics, attendance, completion, follow-up rates, focus groups data and interviews of those who drop out. Evaluation of effect size included the patterns of growth over 15 months from baseline in relation to expected growth patterns and intervention exposure.

ELIGIBILITY:
Inclusion Criteria:

* Children in the 3rd to 5th grades and above the 85th percentile of BMI for age.

Exclusion Criteria:

* Conditions that would preclude dietary change or physical activity.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
body mass index age-and-gender specific Z-score | 9 months post intervention baseline
  body mass index is weight over height squared; z-score described the position of that BMI in relation to the reference population in terms of standard deviation units. It is used to control for growth effects in children.

SECONDARY OUTCOMES:
weight for age-and-gender specific Z-score | 9 months post-intervention baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl K Ritenbaugh, PhD, MPH, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States